CLINICAL TRIAL: NCT07143461
Title: The Effects of Prayer on Pain Thresholds and Scores of Anxiety and Depression in Patients With Migraine and Control: a Randomized Clinical Trial
Brief Title: The Effects of Prayer on Pain Thresholds and Scores of Anxiety and Depression in Patients With Migraine and Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Georgia Kleinschmitt Westenhofen, Sub-Investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1316-9878
Record Dates: First submitted 2025-07-01; First posted 2025-08-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Faith Healing

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized crossover trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researcher will not know which intervention was performed on the first and last day until the study is completed. Randomization will be conducted using two envelopes, each containing the description of one of the two interventions: prayer or reading the control text for 10 minutes. During the first assessment, the envelope chosen by the participant will indicate the procedure to be performed. During the second assessment (follow-up), the remaining intervention (the one not performed on the first day) will be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Migraine + prayer (Experimental): Each migraine participant will serve as their own control, meaning they will undergo both the prayer intervention and the control text intervention on different days. This arm is for the migraine participant and the prayer intervention.
  Interventions: Behavioral: Faith Healing
- Migraine + control text reading (Active Comparator): Each migraine participant will serve as their own control, meaning they will undergo both the prayer intervention and the control text intervention on different days. This arm is for the migraine participant and the control text reading intervention.
  Interventions: Behavioral: Control
- Non-migraine + prayer (Experimental): Each non-migraine participant will serve as their own control, meaning they will undergo both the prayer intervention and the control text intervention on different days. This arm is for the migraine participant and the prayer intervention.
  Interventions: Behavioral: Faith Healing
- Non-migraine + control text reading (Active Comparator): Each non-migraine participant will serve as their own control, meaning they will undergo both the prayer intervention and the control text intervention on different days. This arm is for the migraine participant and the control text reading intervention.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Faith Healing — In the prayer condition, the participants will engage and vocalize in prayers they are already familiar with and commonly practice at least once, then continue silently for 10 minutes, focusing on the content. If distracted, participants should refocus on the prayer and reflect on its meaning.
  Arms: Migraine + prayer; Non-migraine + prayer
Behavioral: Control — In the control condition, participants will read a neutral text with no spiritual or religious content for 10 minutes. If distracted, they should refocus on the text.
  Arms: Migraine + control text reading; Non-migraine + control text reading

SUMMARY:
The objective of this randomized single-blind crossover study is to evaluate the effect of prayer compared to the practice of reading a text (control) on the pressure pain threshold in individuals with and without migraine. The main topics it aims to answer are:

* To analyze the relationship between individuals' spirituality, pain thresholds, and anxiety and depression scores.
* To evaluate the effects of different aspects of prayer (thanksgiving, adoration, confession, meditative, and petitionary) on cephalic pain thresholds in individuals with and without migraines.

Migraine group: 50 participants. Non-migraine group: 50 participants. Total number of participants in total: 100.

DETAILED DESCRIPTION:
Pressure pain thresholds (PPT) represent each person's sensitivity, where the pressure is gradually increased, and participants report when the applied pressure changes from a sensation of pressure to a sensation of pressure and pain. The NOD device is equipped with a digital algometry function, providing reliable quantification of the pressure pain threshold for each individual. For proper use, a 1 cm² adapter will be attached to the front of the device. The tip of this adapter will be positioned perpendicularly to the anatomical structures to be assessed: the temporal region, frontal region, occipital nerve, and vertex. Pain threshold, defined as the minimum pressure required to provoke pain, will be measured in Kg/cm².

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic or episodic migraine.
* Feeling comfortable performing a known prayer.

Exclusion Criteria:

* Severe acute circulatory disorders
* Decompensated diabetes mellitus
* Cognitive weaknesses that prevent the patient from understanding and carrying out the study procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Prayer and pressure pain threshold in Kilopascal (kPa) | Immediately after the intervention session
  To evaluate the effect of prayer compared to the practice of reading a text (control) on the pressure pain threshold in kilopascal unit (kPa) in individuals with and without migraine. To assess the pressure pain threshold, a digital algometer will be used, which measures pain tolerance in kilopascals (kPa).

SECONDARY OUTCOMES:
Spirituality scores using the Functional Assessment of Chronic Illness Therapy - Spiritual Well-being (FACIT-Sp) scale | Immediately after the intervention session
  The FACIT-Sp scale assesses the spiritual well-being of volunteers, focusing on the existential aspects of spirituality and faith. It consists of 12 statements, which are rated on a scale ranging from "not at all," "a little," "somewhat," "quite a bit," to "very much." Higher scores indicate a higher level of spirituality. This assessment does not presuppose belief in God, and therefore does not limit the ability of atheists and agnostics to respond.
Level of religiosity using the Duke Religious Index (DUREL) | Immediately after the intervention session
  To collect data on religiosity, the Duke Religious Index (DUREL) was used to assess the participants' religious involvement. The scale includes five items that address three dimensions of religiosity directly related to health outcomes: organizational religious activity (ORA), non-organizational religious activity (NORA), and intrinsic religiosity (IR). In the validated Portuguese version, lower scores indicate higher levels of religiosity.
Anxiety Variables using Generalized Anxiety Disorder Screener (GAD-7 Scale) | Immediately after the intervention session
  The Generalized Anxiety Disorder Screener (GAD-7) is a 7-item tool based on DSM-IV criteria. It is a unidimensional and easy-to-administer scale designed to assess the presence of generalized anxiety disorder (GAD) symptoms. Each of the 7 items is scored from 0 (not at all) to 3 (nearly every day), resulting in a total score ranging from 0 to 21. The scores are categorized into four severity levels: minimal/no anxiety (0-4), mild (5-9), moderate (10-14), and severe (15-21).
Depression Variables - Patient Health Questionnaire (PHQ-9 Scale) | Immediately after the intervention session
  To identify individuals at risk of depression there is the Patient Health Questionnaire-9 (PHQ-9), a scale based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). It consists of nine items that assess different symptoms. The frequency of each symptom over the past two weeks is rated on a Likert scale from 0 to 3, corresponding to the responses "not at all," "several days," "more than half the days," and "nearly every day," respectively. The higher the score, the greater the levels of depressive symptoms.

OTHER OUTCOMES:
Different aspects of prayer on the pressure pain threshold in Kilopascal (kPa) | Immediately after the intervention session
  To evaluate the effects of different aspects of prayer (thanksgiving, adoration, confession, meditative, and petitionary) on cephalic pressure pain thresholds in individuals with and without migraines. To assess the pressure pain threshold, a digital algometer will be used, which measures pain tolerance in kilopascals (kPa).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry of the University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No